CLINICAL TRIAL: NCT01644149
Title: A Randomized Controlled Clinical Trial Assessing the Immunologic Response to an FDA-approved Influenza Vaccine Delivered Using an FDA-Cleared Jet Injection Vaccine Delivery Device or a Needle and Syringe
Brief Title: Clinical Trial Assessing the Immunologic Response to a Influenza Vaccine Delivered Using an Jet Injection Device or a Needle Syringe
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PharmaJet, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PJ-500-07
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Results first posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Influenza Prophylaxis
Keywords: Jet Injector; Stratis®; PharmaJet; Jet Injection
MeSH Terms: interventions — Needles; Syringes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stratis Jet Injector (Experimental): Single intramuscular administration of 0.5 mL of 2011-2012 Fluzone trivalent inactivated influenza vaccine using the Stratis Jet Injector
  Interventions: Device: Stratis Jet Injector; Biological: 2011-2012 Fluzone trivalent inactivated influenza vaccine
- Needle and Syringe (Active Comparator): Single intramuscular administration of 0.5 mL of 2011-2012 Fluzone trivalent inactivated influenza vaccine using Needle and Syringe
  Interventions: Device: Needle and Syringe; Biological: 2011-2012 Fluzone trivalent inactivated influenza vaccine

INTERVENTIONS:
Device: Stratis Jet Injector — Intramuscular administration of 0.5 mL of 2011-2012 Fluzone trivalent inactivated influenza vaccine
  Other Names: Jet Injector; Disposable Syringe Jet Injector; DSJI
  Arms: Stratis Jet Injector
Device: Needle and Syringe — Intramuscular administration of 0.5 mL of 2011-2012 Fluzone trivalent inactivated influenza vaccine
  Arms: Needle and Syringe
Biological: 2011-2012 Fluzone trivalent inactivated influenza vaccine

SUMMARY:
The primary objective of this study was to evaluate if administration of a seasonal flu vaccine using a jet injector device is comparable to traditional needle and syringe delivery for eliciting an immune response. A secondary objective was to compare the safety of the two delivery methods.

DETAILED DESCRIPTION:
Needle-free jet injection devices create a fine stream of pressurized liquid that is able to deliver vaccines and other pharmaceutical products beneath the skin. Design aspects such as quality, pressure, orifice size, angle of injection relative to skin and injection stream coherence control the depth to which the product is delivered. This technology provides a safer delivery option for patients and healthcare staff by removing the need for needles for the administration of vaccines.

In addition to improved safety, additional benefits of using jet injectors include more consistent and reliable dose volume delivery, reduced vaccine waste, diminished need to transport large quantities of sharps, reduced risk of needle sticks, syringe reuse, and costs associated with sharps waste. Jet injectors offer a needle-free procedure to those individuals who are adverse to needles.

This study compared the efficacy of a disposable syringe jet injection device (Stratis) with traditional needle and syringe (NS) administration for the delivery of a trivalent inactivated influenza vaccine. Efficacy was evaluated by comparing measures of hemagglutination inhibition (HI); specifically GMTs, seroconversion and seroprotection. Safety of the two administration devices was evaluated by comparison of incidence of solicited local and systemic adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Female and male subjects ages 18 to 59 years
* Healthy volunteers
* Able to provide informed consent and understand study procedures per ICH/GCP guidelines
* Plans to remain in study area for length of the trial; able to adhere to study visit and follow-up schedule
* Able to complete study diary

Exclusion Criteria:

* Unwilling or unable to undergo the two blood draws per protocol
* Have received influenza vaccination in the last twelve months
* Have received any vaccination in the last month
* Currently taking antibiotics, steroids, phenytoin, chemotherapy, or other immunosuppressive drugs
* Received recent blood, blood products, or parenteral preparations of immunoglobulin (within 3 months)
* Suffers from allergic reactions to egg, gelatin, or neomycin or has a history of anaphylactic shock, asthma, urticaria, or other allergic reactions to vaccinations.
* Had any serious adverse event associated with a prior vaccination
* Has immunodeficiency or autoimmune disease (including HIV)
* History of chronic alcohol abuse
* Participating in another study concurrently
* Pregnant or breastfeeding during the study

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2012-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Perlman, MD, MBA, Principal Investigator — Bel-Rea Institute
Locations (1):
- Bel-Rea Institute, Denver, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Up to 100 subjects between the ages of 18 and 59 were planned with 83 subjects enrolled and 82 subjects vaccinated. Pre- and post-vaccination serum samples were collected from 78 subjects and were analyzed in the Efficacy population.
Pre-assignment Details: A total of 83 subjects were recruited and 78 (39 Stratis® and 39 NS) completed the study. One Stratis® group subject (subject # 23) discontinued from the study prior to vaccination.
Groups:
- Stratis Jet Injector: Patients assigned to this arm will receive Fluzone trivalent inactivated influenza vaccine administered using the STRATIS needle-free injection device. Fluzone vaccine (2011-2012 formulation): Patients will receive a single intramuscular injection of 0.5 ml of Fluzone vaccine in the deltoid region.
  STRATIS needle-free injection device
- Needle-Syringe: Patients assigned to this arm will receive Fluzone trivalent inactivated influenza vaccine administered using a needle and syringe. Fluzone vaccine (2011-2012 formulation): Patients will receive a single intramuscular injection of 0.5 ml of Fluzone vaccine in the deltoid region.
  Needle-Syringe
Period: Overall Study
Arm/Group | Stratis Jet Injector | Needle-Syringe
Started | 43 | 40
Completed | 39 (One subject discontinued prior to vaccination. 28 day serum samples not obtained from 3 subjects.) | 39 (28 day serum samples were not obtained from one NS subject.)
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- PharmaJet Stratis Injector: Single intramuscular administration of 0.5 mL of 2011-2012 Fluzone trivalent inactivated influenza vaccine using the Stratis Jet Injector
  Stratis Jet Injector: Intramuscular administration of 0.5 mL of 2011-2012 Fluzone trivalent inactivated influenza vaccine
  2011-2012 Fluzone trivalent inactivated influenza vaccine
- Needle and Syringe: Single intramuscular administration of 0.5 mL of 2011-2012 Fluzone trivalent inactivated influenza vaccine using Needle and Syringe
  Needle and Syringe: Intramuscular administration of 0.5 mL of 2011-2012 Fluzone trivalent inactivated influenza vaccine
  2011-2012 Fluzone trivalent inactivated influenza vaccine
- Total: Total of all reporting groups
Arm/Group | PharmaJet Stratis Injector | Needle and Syringe | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 39 | 78
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 26 | 54
  Male | 11 | 13 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 34 | 31 | 65
  Asian | 1 | 2 | 3
  Black or African American | 1 | 1 | 2
  Hispanic or Latino | 2 | 4 | 6
  American Indian or Alaska Native | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 39 | 39 | 78

OUTCOME MEASURES:

1. Primary Outcome: Anti Influenza Hemagglutination Inhibition (HAI) Antibody Geometric Mean Titers (GMT)
Description: The GMT criterion for non-inferiority for the upper limit of the 95% CIs of the GMT ratio (GMT with Needle-Free / GMT with Needle and Syringe) antigen will not exceed 1.5 fold.
Time Frame: 28 days
Population: The immunogenicity analyses were conducted using data from subjects in the immunogenicity population.
Measure: Geometric Mean (Standard Deviation); unit: Titers
Groups:
- Stratis Jet Injector: Patients assigned to this arm will receive Fluzone vaccine administered using the PharmaJet (PJ) STRATIS needle-free injection device.
  Fluzone vaccine (2011-2012 formulation): Patients will receive a single 0.5 mL injection of Fluzone vaccine in the deltoid region.
  PJ STRATIS needle-free injection device
- Needle and Syringe: Patients assigned to this arm will receive Fluzone vaccine administered using needle and syringe.
  Fluzone vaccine (2011-2012 formulation): Patients will receive a single 0.5 mL injection of Fluzone vaccine in the deltoid region.
  Needle-Syringe.
Arm/Group | Stratis Jet Injector | Needle and Syringe
Number analyzed (Participants) | 39 | 39
Titers
  A/ H1N1 Day 0 | 3.55 (1.19) | 3.49 (1.28)
  A H1N1 Day 28 | 6.19 (0.98) | 6.13 (1.05)
  A/ H3N2 Day 0 | 3.55 (1.30) | 3.49 (1.40)
  A/H3N2 Day 28 | 6.31 (1.28) | 6.14 (1.16)
  B Day 0 | 2.57 (0.51) | 2.53 (0.45)
  B Day 28 | 4.17 (1.00) | 4.17 (1.10)

2. Primary Outcome: The Percentage of Participants Achieving Seroconversion
Description: Seroconversion is defined as a 4-fold rise in HAI titer in post-immunization serum relative to pre-immunization serum, or if pre-immunization serum had an undetectable titer (<1:10), attainment of a post-immunization titer of ≥1:40.
Time Frame: 28 days
Population: Seroconversion against the hemagglutinin antigens contained in the vaccine were assessed in the Immunogenicity Population.
Measure: Number; unit: Percentage of Subjects Seroconverted
Groups:
- Stratis Jet Injector: Patients assigned to this arm will receive Fluzone vaccine administered using the PJ STRATIS needle-free injection device.
  Fluzone vaccine (2011-2012 formulation): Patients will receive a single 0.5 mL injection of Fluzone vaccine in the deltoid region.
  PJ STRATIS needle-free injection device
Arm/Group | Stratis Jet Injector | Needle and Syringe
Number analyzed (Participants) | 39 | 39
Percentage of Subjects Seroconverted
  A/H1N1 | 79.5 | 85.0
  A/H3N2 | 89.7 | 85.0
  B | 59.0 | 65.0

3. Secondary Outcome: Percentage of Subjects With Solicited Local or Systemic Adverse Events
Description: Vaccine reactogenicity will be collected on a patient-completed diary card daily for seven days post-vaccination. The following adverse events will be solicited on the diary card: injection site tenderness, injection site pain, injection site redness, injection site swelling, injection site itching, injection site bruising, fatigue, muscle aches, headache, decreased appetite, fever, pruritus.
Time Frame: 4 days
Population: Data included in the analysis were collected on a 4-Day Diary Card from the safety population and grade >1.
Measure: Number; unit: Percentage of Subjects
Arm/Group | Stratis Jet Injector | Needle and Syringe
Number analyzed (Participants) | 39 | 39
Percentage of Subjects
  Tenderness | 95 | 80
  Pain | 68 | 58
  Redness | 61 | 25
  Swelling | 50 | 20
  Itching | 34 | 13
  Bruising | 26 | 20
  Fatigue | 34 | 38
  Muscle Aches | 47 | 33
  Headache | 34 | 28
  Decreased Appetite | 16 | 20
  Fever | 16 | 18
  Pruritis | 24 | 10

ADVERSE EVENTS:
Time Frame: Complaints were solicited from subjects in the safety population following vaccination: pain, tenderness, itching, redness, swelling, and bruising at the vaccination site. Local and systemic study injection reactions were monitored for 4 days post injection.
Description: Solicited adverse events were those events specifically sought for and recorded by the subject in the 4-Day Diary Card.
  The denominators were determined for each individual AE for each summary window (Day 0-4). Subjects in Safety Populations were excluded from the denominator if there was no data captured for the AE within summary window.
Arm/Group | PharmaJet Stratis Injector | Needle and Syringe
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 36/39 | 32/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PharmaJet Stratis Injector (N=39) | Needle and Syringe (N=39)
Tenderness (General disorders) | 36 | 32 — Local Adverse Reaction within 4 days of vaccination and Grade of >=1
Pain (General disorders) | 26 | 23 — Local symptoms at injection site within 4 days of vaccination with Grade of >=1
Redness (General disorders) | 23 | 10 — Local event occurring within 4 days of vaccination and Grade of >=1
Swelling (General disorders) | 19 | 8 — Local event occurring within 4 days of vaccination and Grade of >=1
Itching (General disorders) | 13 | 5 — Local event occurring within 4 days of vaccination and Grade of >=1
Bruising (General disorders) | 10 | 8 — Local event occurring within 4 days of vaccination and Grade of >=1
Fatigue (Immune system disorders) | 13 | 15
Muscle Aches (Musculoskeletal and connective tissue disorders) | 18 | 13
Headache (Nervous system disorders) | 13 | 11
Decreased Appetite (Gastrointestinal disorders) | 6 | 8
Fever (Nervous system disorders) | 6 | 7
Pruritis (Skin and subcutaneous tissue disorders) | 9 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less